CLINICAL TRIAL: NCT06067841
Title: A Phase 1, Open-label Study of BMS-986460 in Participants With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study to Assess BMS-986460 in Participants With Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA125-1008; 2024-513987-24 (Other: EU CTR); U1111-1307-2450 (Other: WHO)
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate Cancer; Castration-resistant prostate cancer; Adenocarcinoma of the prostate; Prostatic Neoplasms Castration-Resistant; Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of BMS-986460 (Experimental)
  Interventions: Drug: BMS-986460

INTERVENTIONS:
Drug: BMS-986460 — Specified dose on specified days.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and preliminary efficacy of BMS-986460 in men with Metastatic Castration-resistant Prostate Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed adenocarcinoma of the prostate.
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Participant must have prostate specific antigen (PSA) of ≥ 2 ng/mL at Screening
* Participant must have progressed on androgen deprivation therapy (ADT) and at least one prior secondary hormonal therapy approved for castration-resistant prostate cancer (CRPC)

Exclusion Criteria:

* Participant must not have history of brain metastases.
* Participant must not have impaired cardiac function or clinically significant cardiac disease.
* Participant must not have any significant medical condition, including active or uncontrolled infection, psychiatric illness, or the presence of laboratory abnormalities, which places the participant at unacceptable risk or prevent participation in the study based on Investigator assessment.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2029-08-24 (Estimated); Study Completion 2031-07-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 112 weeks
Number of participants with serious adverse events (SAEs) | Up to 112 weeks
Number of participants with AEs meeting protocol defined dose limiting toxicity (DLT) criteria | Up to 28 days
Number of participants with AEs leading to study intervention discontinuation | Up to 104 weeks
Number of deaths | Up to 108 weeks

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Up to 13 weeks
Time of maximum concentration (Tmax) | Up to 13 weeks
Area under the plasma concentration-time curve (AUC) | Up to 13 weeks
Number of participants with a confirmed prostate specific antigen decline of ≥ 30% from baseline response rate | Up to 108 weeks
Number of participants with soft tissue response | Up to 108 weeks
Duration of response (DOR) | Up to 108 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (8):
  - Stanford Cancer Center, Palo Alto, California
  - Florida Cancer Specialists Sarasota Drug Development Unit, Sarasota, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Local Institution - 0006, San Antonio, Texas
  - NEXT Oncology, San Antonio, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06067841.html